CLINICAL TRIAL: NCT01440309
Title: Phase I Clinical Trial, Randomized, Controlled, to Evaluate the Efficacy and Safety of Therapy With Allogenic Mesenchymal Stem Cells From Bone Marrow for Patients With Refractory Primary Biliary Cirrhosis
Brief Title: Efficacy and Safety Study of Allogenic Mesenchymal Stem Cells for Patients With Refractory Primary Biliary Cirrhosis
Acronym: MSCsTreatPBC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Robert Chunhua Zhao, MD, PhD (Unknown)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Robert Chunhua Zhao, MD, PhD, MD, PhD，Professor of medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008BAI59B03/2011AA020119
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2011-09

CONDITIONS: Primary Biliary Cirrhosis
Keywords: biliary cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allogenic mesenchymal stem cells (MSCs) (Experimental): Patients who have primary biliary cirrhosis.
  Interventions: Biological: Biological: mesenchymal stem cell
- ursodeoxycholic acid (UDCA) (Active Comparator): Patients who have primary biliary cirrhosis.
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Biological: Biological: mesenchymal stem cell — Mesenchymal stem cells,5-50 million/kg, Intravenous infusion, One dosage，whether to give another dosage depending on patients' condition
  Other Names: regenerative medicine:MSCs
  Arms: allogenic mesenchymal stem cells (MSCs)
Drug: ursodeoxycholic acid — 13-15 mg/kg/day, to the end of the study
  Other Names: UDCA
  Arms: ursodeoxycholic acid (UDCA)

SUMMARY:
The study is designed to evaluate the safety and efficacy of intravenous administration of bone marrow derived mesenchymal stem cells for patients with refractory primary biliary cirrhosis (PBC).

DETAILED DESCRIPTION:
Primary biliary cirrhosis (PBC) is an organ-specific inflammatory disease and characterized by immune mediated destruction of intrahepatic bile ducts, then lead to liver cirrhosis and eventually failure.Currently, ursodeoxycholic acid (UDCA) is the only drug approved by the Food and Drug Administration (FDA). Novel treatment is urgently needed for patients who have an incomplete response to UDCA. Mesenchymal stem cells (MSC) represent a promising tool for cell-based therapies of autoimmune diseases. To explore the therapeutic effect of MSCs for PBC, the investigators plan to conduct an open-label, randomized clinical trial. Patients with PBC will be enrolled and randomly divided into two groups which will receive MSCs and UDCA respectively. The investigators will evaluate the efficacy and safety of MSCs for PBC by comparison of symptom improvement, survival rate and side effects in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* There must be at least two of the following: a concentration in serum of AMAs at titres of 1:40 or higher; an unexplained rise in the amount of alkaline phosphatase of at least 1•5 times the upper limit of normal for more than 24 weeks; and compatible liver histological findings, specifically non-suppurative cholangitis and interlobular bile duct injury.
* Incomplete response to UDCA at 13-15 mg/kg/day, Criteria for the group of complete responders is including: concentrations of alkaline phosphatase less than three times the upper limit of normal, aspartate aminotransferase less than twice the upper limit of normal, and bilirubin less than 17 μmol/L;and normalisation of abnormal concentrations of bilirubin, albumin, or both.
* Liver pathological staging in 2 or3, Histological staging is based on Ludwig's and Scheuer's classifications

Exclusion Criteria:

* Patients are receiving any other investigational agents within 4 weeks of study entry
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined as invasive fungal infection and progressive CMV viremia), symptomatic congestive heart failure (NYH class III and IV), unstable angina pectoris, or cardiac arrhythmia
* In pregnancy or lactation
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
* HCVpositive ，HBSAg positive or with other liver diseases
* Combined with other autoimmune disease
* Expected survival time is less than one year
* Decompensation of liver function（Child B or C）
* Have a history of allergy or Allergic constitution

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
serum level of alkaline phosphatase | 24 months after MSCs administration
  Serum level of alkaline phosphatase will be measured at entry, 1 months，3 months, 6 months and 24 months after therapy

SECONDARY OUTCOMES:
histological changes in liver biopsies | 6 months after therapy
  Liver biopsy of each patient will be taken before entry into therapeutic trials and at 6 months after therapy.
Serum levels of TNF-alpha | 6 months after therapy
  serum levels of TNF-alpha will be assessed before entry into therapeutic trials and at 6 months after therapy
changes in fatigue | 6 months after theraphy
  changes in fatigue will be evaluated before test (baseline), 1 month,3 months and 6 months after theraphy by PBC-40 score.
The occurrence of cirrhosis and its complications | 24 months after therapy
Serum levels of Interleukin | 6 months after therapy
  serum levels of Interleukin will be assessed before entry into therapeutic trials and at 6 months after therapy
changes in pruritus severity | 6 months after therapy
  changes in pruritus severity will be evaluated before test (baseline), 1 month,3 months and 6 months after theraphy by VAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, MD, Principal Investigator — Peking Union Medical College Hospital; Robert Chunhua Zhao, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Background] Sun Z, Han Q, Zhu Y, Li Z, Chen B, Liao L, Bian C, Li J, Shao C, Zhao RC. NANOG has a role in mesenchymal stem cells' immunomodulatory effect. Stem Cells Dev. 2011 Sep;20(9):1521-8. doi: 10.1089/scd.2010.0366. Epub 2011 Feb 26. PMID 21235326
- [Background] Shi D, Liao L, Zhang B, Liu R, Dou X, Li J, Zhu X, Yu L, Chen D, Zhao RC. Human adipose tissue-derived mesenchymal stem cells facilitate the immunosuppressive effect of cyclosporin A on T lymphocytes through Jagged-1-mediated inhibition of NF-kappaB signaling. Exp Hematol. 2011 Feb;39(2):214-224.e1. doi: 10.1016/j.exphem.2010.10.009. Epub 2010 Nov 13. PMID 21078360
- [Background] Zhang B, Liu R, Shi D, Liu X, Chen Y, Dou X, Zhu X, Lu C, Liang W, Liao L, Zenke M, Zhao RC. Mesenchymal stem cells induce mature dendritic cells into a novel Jagged-2-dependent regulatory dendritic cell population. Blood. 2009 Jan 1;113(1):46-57. doi: 10.1182/blood-2008-04-154138. Epub 2008 Oct 2. PMID 18832657
- [Background] Liao L, Zhao RC. An overview of stem cell-based clinical trials in China. Stem Cells Dev. 2008 Aug;17(4):613-8. doi: 10.1089/scd.2008.0183. PMID 18673001
- [Background] Fang B, Shi M, Liao L, Yang S, Liu Y, Zhao RC. Systemic infusion of FLK1(+) mesenchymal stem cells ameliorate carbon tetrachloride-induced liver fibrosis in mice. Transplantation. 2004 Jul 15;78(1):83-8. doi: 10.1097/01.tp.0000128326.95294.14. PMID 15257043
- [Background] Wang J, Bian C, Liao L, Zhu Y, Li J, Zeng L, Zhao RC. Inhibition of hepatic stellate cells proliferation by mesenchymal stem cells and the possible mechanisms. Hepatol Res. 2009 Dec;39(12):1219-28. doi: 10.1111/j.1872-034X.2009.00564.x. Epub 2009 Sep 25. PMID 19788697
- [Background] Chen L, Zhang W, Yue H, Han Q, Chen B, Shi M, Li J, Li B, You S, Shi Y, Zhao RC. Effects of human mesenchymal stem cells on the differentiation of dendritic cells from CD34+ cells. Stem Cells Dev. 2007 Oct;16(5):719-31. doi: 10.1089/scd.2007.0065. PMID 17999594
- [Background] Deng W, Han Q, Liao L, You S, Deng H, Zhao RC. Effects of allogeneic bone marrow-derived mesenchymal stem cells on T and B lymphocytes from BXSB mice. DNA Cell Biol. 2005 Jul;24(7):458-63. doi: 10.1089/dna.2005.24.458. PMID 16008514
- [Background] Deng W, Han Q, Liao L, Li C, Ge W, Zhao Z, You S, Deng H, Zhao RC. Allogeneic bone marrow-derived flk-1+Sca-1- mesenchymal stem cells leads to stable mixed chimerism and donor-specific tolerance. Exp Hematol. 2004 Sep;32(9):861-7. doi: 10.1016/j.exphem.2004.06.009. PMID 15345288
- [Background] Zhang W, Ge W, Li C, You S, Liao L, Han Q, Deng W, Zhao RC. Effects of mesenchymal stem cells on differentiation, maturation, and function of human monocyte-derived dendritic cells. Stem Cells Dev. 2004 Jun;13(3):263-71. doi: 10.1089/154732804323099190. PMID 15186722